CLINICAL TRIAL: NCT04699656
Title: A Phase 1 Open-Label Study to Assess the Pharmacokinetics, Safety, and Tolerability of Intravenous Administration of Plazomicin in Subjects With End Stage Renal Disease (ESRD) Receiving Intermittent Hemodialysis (IHD)
Brief Title: Plazomicin Study in ESRD Patients Receiving IHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cipla USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPH-002-CL-013
Record Dates: First submitted 2020-12-28; First posted 2021-01-07 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — plazomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Plazomicin Injection (Experimental): plazomicin (30-minute IV infusion at 2.5 mg/kg) single dose given before IHD and single dose given after IHD
  Interventions: Drug: Plazomicin Injection

INTERVENTIONS:
Drug: Plazomicin Injection — single dose of plazomicin
  Other Names: Zemdri

SUMMARY:
This study is being conducted to directly characterize the pharmacokinetic (PK) profile of plazomicin following administration of a single oral dose before and after IHD in subjects with ESRD. This PK assessment will be used to provide appropriate plazomicin dosing recommendations for patients with ESRD receiving IHD.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label, single-dose study to evaluate the PK of a single dose of plazomicin (30-minute IV infusion at 2.5 mg/kg) when administered prior to and after IHD in subjects with ESRD.

The study will consist of a screening period of up to 28 days and two treatment periods, with at least a 7-day washout between dosing in each treatment period. The start of the study is defined as the date that the first subject is screened following signing of an informed consent form (ICF).

In Period 1 (Week 1), the dosing day will be concomitant with the 3rd weekly IHD session, which must be at least 72 hours before the 1st weekly IHD session of the subsequent Week. All subjects will receive a single dose of plazomicin (30 minute IV infusion at 2.5 mg/kg) within 1 hour after IHD is completed. PK samples will be collected at specified time points from 0.6 hours to 72 hours after completion of the plazomicin infusion. Collection of all PK samples must be completed prior to the next scheduled IHD.

In Period 2 (Week 2), the dosing day will occur on the day of the 3rd weekly IHD session, which must be at least 7 days after the first dose and at least 72 hours before the 1st weekly IHD session of the subsequent Week. All subjects will receive a single dose of plazomicin (30 minute IV infusion at 2.5 mg/kg) before IHD is started. The plazomicin infusion should be completed within 30 minutes of IHD initiation. During IHD, the total dialysate will be collected in a large collection container and pooled at 1-hour intervals (0-1, 1-2, 2-3, etc. for the duration of the IHD session). From each hourly interval (including any partial interval at end of dialysis), an aliquot sample of dialysate will be collected for PK analysis. PK samples will be collected at specified time points from 0.6 hours to 72 hours after completion of the plazomicin infusion. Collection of all PK samples must be completed prior to the next scheduled IHD.

Safety assessments will include physical examination findings, vital signs (blood pressure, pulse rate, respiration rate, and oral temperature), clinical laboratory evaluations, and monitoring of adverse events (AEs). Adverse events will be assessed from the time the subject signs the ICF until exit from the study.

The site will attempt to contact all subjects (including subjects who terminate the study early) via phone call approximately 14 days after the last dose of study drug to determine if any AE has occurred since the last study visit. Subjects reporting AEs may be asked to return to the site for further assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 75 years of age with a BMI ≥19 to ≤42 kg/m2 and weight of ≥40 kg
* Pre-existing ESRD requiring in-center IHD for a minimum of 3 months on a schedule of three IHD sessions per week with the third weekly IHD session occurring at least 72 hours before the first weekly IHD session of the subsequent week (e.g. Monday/Wednesday/Friday or Tuesday/Thursday/Saturday)
* Females of childbearing potential must not be breast-feeding, must have a negative serum pregnancy test at screening, and must use a highly effective method of contraception (includes hormonal implants, intrauterine devices, injectable hormones, oral hormonal contraceptives, prior hysterectomy, prior bilateral oophorectomy, or a vasectomized partner whose vasectomy was performed 4 months or more prior to dosing on Day 1) or be abstinent from sexual activity for at least 1 month prior to dosing on Day 1, during the study and through 30 days following the last dose of study drug. Females of non-childbearing potential, defined as women who have not had a period for 12 consecutive months prior to dosing on Day 1, may be enrolled.
* Willing to comply with all study activities and procedures and have provided written informed consent prior to any study procedures and have signed and dated a Health Insurance Portability and Accountability Act (HIPAA) authorization form.

Exclusion Criteria:

* Subjects with any medical, psychological, or social condition which, in the opinion of the Investigator, would prevent the subject from fully participating in the study, would represent a concern for study compliance or would constitute a safety concern to the subject.
* Unstable cardiovascular disease per the Investigator, including:

  1. Heart rate <40 or >110 beats per minute (bpm) or QT interval corrected using Fridericia's formula (QTcF) >500 msec.
  2. Uncontrolled hypertension, asthma, diabetes (type I or type II), thyroid disease, or seizure disorder
* Myasthenia gravis or any other neuromuscular disorder.
* Known infection with hepatitis B (antigen positive), hepatitis C (antibody positive), or human immunodeficiency virus (HIV). Subjects with clinically insignificant or adequately treated hepatitis C may be allowed at the discretion of the Investigator.
* Active malignancy; carcinoma in situ of the prostate or cervix or basal cell or squamous cell carcinoma of the skin are permitted.
* Presence of functioning transplant organ or blood procedure.
* Significant change in either over-the-counter or prescription medications or supplements within 3 months prior to dosing, defined as any new medication or any dosage adjustment that is significant in the judgment of the Investigator.
* History of significant hearing loss or a family history of hearing loss, excluding age-related (≥65 years) hearing loss. A prior diagnosis of sensorineural hearing loss or Ménière's disease or receipt of any potentially ototoxic agent within 30 prior to the start of screening.
* Subjects who received a systemic aminoglycoside within 90 days of the start of screening.
* Clinically significant illness, including viral syndromes within three weeks of dosing.
* Current participation in a clinical study of an investigational product.
* Subjects who took any investigational medication/therapy within 30 days or 5 half-lives, whichever is longer, before dosing of plazomicin.
* Subjects with active alcoholism and/or drug/chemical abuse in the opinion of the Investigator. Also, consumption of any amount of ethanol within 48 hours of plazomicin dosing.
* Subjects who donated more than 500 mL of blood within 60 days prior to start of screening.
* Previous participation in this or any other plazomicin study.
* Known hypersensitivity to aminoglycosides or any component of plazomicin injection.
* The subject is an employee of the Investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member of the employee or Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
o Maximum observed plasma drug concentration (Cmax) | 30 days
  Plasma PK parameter for plazomicin before and after IHD
o Time to maximum observed plasma concentration (Tmax) | 30 days
  Plasma PK parameter for plazomicin before and after IHD
o Area under the plasma concentration time curve from time 0 to the last measurable concentration (AUC0-t) | 30 days
  Plasma PK parameter for plazomicin before and after IHD
o Area under the plasma concentration time curve extrapolated to infinity (AUCinf) | 30 days
  Plasma PK parameter for plazomicin before and after IHD
o Terminal elimination half-life (t1/2) | 30 days
  Plasma PK parameter for plazomicin before and after IHD
o Total plasma clearance (CL) | 30 days
  Plasma PK parameter for plazomicin before and after IHD
o Volume of distribution during the terminal elimination phase (Vz) | 30 days
  Plasma PK parameter for plazomicin before and after IHD
o Terminal elimination rate constant (λz) | 30 days
  Plasma PK parameter for plazomicin before and after IHD

SECONDARY OUTCOMES:
• Adverse events (AEs) | 30 days
  Safety assessment; An overall summary will be generated presenting the frequency and percentage of subjects and the number of treatment-emergent adverse events (TEAEs).

OTHER OUTCOMES:
o Cumulative amount of drug excreted in dialysate (Ae) | 30 days
  Dialysate PK parameter for plazomicin after IHD
o Percent of plazomicin recovered in dialysate (Ae%) | 30 days
  Dialysate PK parameter for plazomicin after IHD
o Dialysate clearance (CLD) | 30 days
  Dialysate PK parameter for plazomicin after IHD

CONTACTS AND LOCATIONS:
Overall Officials: Patrice P Rioux, MD, PhD, Study Director — Cipla USA Inc.
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States